CLINICAL TRIAL: NCT05510661
Title: Use of Export in Primary Percutaneous Coronary Intervention, In-Hospital and Short-term Outcomes and Optimal Time of Export
Brief Title: Use of Export in Primary Percutaneous Coronary Intervention
Acronym: EPISOO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Faiza Farooq, Acting Associate Professor, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERC-63/2021
Record Dates: First submitted 2021-06-30; First posted 2022-08-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI); Total Occlusion of Coronary Artery; Primary Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Manual thrombus aspiration (use of export catheter) followed by primary PCI
Who Masked: Outcomes Assessor
Masking Description: Blinded in-hospital outcomes assessment will be insured by separating patients recruitment and follow-up team and follow-up team will be kept blinded of randomization. All the patients will be assigned a unique identity code and collected data will be stored against the assigned code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Group (Experimental): Manual thrombus aspiration (use of export catheter) followed by primary PCI
  Interventions: Device: Export Catheter
- Control group (Active Comparator): Predilatation with balloon catheter (≤2.00 mm diameter) followed by primary PCI
  Interventions: Device: Balloon catheter

INTERVENTIONS:
Device: Export Catheter — Manual thrombus aspiration with the use of export catheter during primary PCI
  Other Names: Thrombus Aspiration
  Arms: Intervention Group
Device: Balloon catheter — Predilatation with balloon catheter
  Arms: Control group

SUMMARY:
Aim of this single center randomized open label trial with blinded in-hospital outcomes assessment is designed with aim to compare manual thrombus aspiration followed by percutaneous coronary intervention (PCI) strategy with PCI alone.

DETAILED DESCRIPTION:
Clinical benefit of manual aspiration has been a contentious point of debate and it is Class III indication in current clinical practice guidelines, however, recent observational data by Kumar D et al. showed benefits of usage of export in terms of favorable in-hospital outcomes and lesser complication rate in patients with total occlusion, furthermore, benefits of usage of export was observed to be directly associated with duration of chest pain at the time of thrombus aspiration. However, these observations are limited to immediate and in-hospital outcomes and data regarding efficacy of manual thrombus aspiration are not available.

Hence this single center randomized open label trial is designed with specific aim to test the following hypothesis for STEMI patients with total occlusion undergoing primary PCI;

* Whether use of export catheter reduces in-hospital and short term adverse events
* Whether use of export reduces slow flow or no reflow
* Whether use of export reduces the use of intracoronary drugs
* Whether use of export within 6 hours of symptom onset significantly reduces in-hospital and short term adverse events

Consecutively recruited patients will be randomized to either primary PCI with export or primary PCI alone group in 2:1 ratio. Post aspiration immediate TIMI flow will be observed and all the patients will be observed for adverse outcomes (MACE) and complications including slow flow/no-reflow. Follow-up intervals will be at the end of one month of randomization and end of 6 month of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with:-Symptoms of myocardial ischemia lasting for ≥30 minutes
* Definite ECG changes indicating STEMI: ST elevation of greater than 0.1 mV in two contiguous limb leads or 0.2 mV in two contiguous precordial leads
* Chest pain < 12 hours duration
* Total occlusion (TIMI 0 flow)
* Patients undergoing primary PCI
* Informed consent

Exclusion Criteria:

* Patients with prior history of cardiac related surgery or intervention
* Performance of a rescue PCI after thrombolysis
* Known existence of a disease resulting in a life expectancy of less than 6 months
* Killip class III, IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Post thrombus aspiration TIMI flow | Immediately after export/balloon
  Immediate TIMI flow after export/balloon
Slow/No-reflow | Immediately after procedure
  TIMI 0-II flow
Major adverse cardiac events | In-hospital, at 1 month, and at 6 months
  It will include All-cause death, Cardiovascular death, Re- infarction, Heart Failure, Cardiogenic shock, Cerebrovascular events, Bleeding events, and Stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Dr Fiaza Farooq, FCPS, Principal Investigator — National Institute of Cardiovascular Diseases (NICVD), Karachi, Pakistan
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kumar D, Saghir T, Sial JA, Kumar R, Karim M, Huma ZE, Qamar N. Use of export vs. balloon in primary percutaneous coronary intervention, in-hospital outcomes and optimal export time. Journal of the American College of Cardiology. 2021 May 11; 77(18_Supplement_1): 1034.